CLINICAL TRIAL: NCT02926365
Title: Increased Access to Psychological Treatment for Children and Adolescents Through Internet-delivered CBT - a Pragmatic Evaluation Within Regular Health Care in a Rural Area of Sweden
Brief Title: BIP in Jämtland Härjedalen: Increased Access to CBT Within Regular Health Care in Northern Sweden
Acronym: BIPBJÖRN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sarah Vigerland, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPN DNR 2016/1355-31/5
Record Dates: First submitted 2016-09-20; First posted 2016-10-06 (Estimated); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Anxiety Disorder; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Anxiety Disorders; Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICBT (Experimental): Therapist-supported internet-delivered CBT
  Interventions: Behavioral: ICBT

INTERVENTIONS:
Behavioral: ICBT

SUMMARY:
The purpose of this study is to test internet-delivered cognitive behavior therapy for children and adolescents with anxiety disorders and obsessive-compulsive disorder in a routine clinical setting in a rural part of Sweden.

DETAILED DESCRIPTION:
Aim The aim of this study is to conduct a pragmatic evaluation of ICBT for children and adolescents with anxiety disorders and OCD within routine health care in a rural area.

Research questions

* Is ICBT an acceptable method for the patient group?
* Is ICBT effective in a clinical setting?
* Is further treatment needed after ICBT?
* What are the long-term effects of ICBT?
* What predicts treatment outcome?
* How does ICBT work in a clincal setting? (time spent, negative effects etc)?

Design This is a uncontrolled intervention study where included families and children will be recruited consecutively during two years from a routine care CAMHS unit. All participants will be offered ICBT and assessed pre- and post-treatment, and at three-month follow-up through clinician ratings and self-report measures. The primary outcome measure is clinician rated severity of principal disorder at three-month follow-up. Long-term results will be assessed through study of medical records two years after completed ICBT.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills diagnostic criteria for an anxiety disorder or OCD
* Access to a computer and internet connection
* Read and speak Swedish

Exclusion Criteria:

* ICBT is currently not assessed to be a suitable treatment
* Acute psychiatric problem (eg. severe depression or suicidality)
* Current psychosocial problems in the family (i.e substance abuse, abuse, neglect)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
CGI-S | 24 weeks from baseline
  Clinical Global Impression - Severity

SECONDARY OUTCOMES:
CGI-S | 12 weeks from baseline
  Clinical Global Impression - Severity
CGI-I | 12 and 24 weeks from baseline
  Clinical Global Impression - Improvement
CGAS | 12 and 24 weeks from baseline
  Children's Global Assessment Scale
CY-BOCS | 12 and 24 weeks from baseline
  Children's Yale Brown Obsessive Compulsive Scale
RCADS | 12 and 24 weeks from baseline
  Revised Children's Anxiety and Depression Scale
EWSAS | Week 1 through 12 + 24 weeks from baseline
  Education, Work and Social Adjustment Scale - Child and parent versions
Patient satisfaction | 12 weeks from baseline
  Questionnaire on child- and parent rated treatment satisfaction
Adverse events | 12 weeks from baseline
  Unintended treatment effects - child and parent version

CONTACTS AND LOCATIONS:
Overall Officials: Eva Serlachius, Med Dr, Principal Investigator — Karolinska Institutet
Locations (1):
- BUP Jämtland Härjedalen, Östersund, Region Jämtland Härjedalen, Sweden

IPD SHARING:
Plan to Share IPD: No
No such plan exists at the moment

REFERENCES:
- [Background] Vigerland S, Fredlander S, Aspvall K, Jolstedt M, Lenhard F, Mataix-Cols D, Ljotsson B, Serlachius E. Effectiveness of internet-delivered cognitive behavioural therapy for anxiety and obsessive-compulsive disorders within routine clinical care in rural Sweden. Internet Interv. 2024 Apr 6;36:100738. doi: 10.1016/j.invent.2024.100738. eCollection 2024 Jun. PMID 38617387